# Informed Consent Form

Official Title: Application Research of a Blended Teaching Model Based on Generative Artificial Intelligence in the Practical Teaching of Internal Medicine Nursing

NCT Number: Pending

Document Date: September 13, 2025

Researcher: Wang Hengxu, Senior Nurse

Research Unit: School of Nursing, Changsha Medical University Contact Information: 15575503185 | 1543980936@qq.com

## Dear Nursing Student,

Hello! We sincerely invite you to participate in a teaching reform research project. This study aims to explore new teaching methods to improve the teaching quality of the Internal Medicine Nursing practical course. Before you decide whether to participate, please read the following content carefully to fully understand the purpose, procedures, potential benefits, risks, and your rights and obligations regarding this research. If you have any questions, please feel free to ask us at any time.

# 1. Research Purpose and Background

This study aims to develop and test a blended online and offline teaching model that integrates generative artificial intelligence (AI), virtual simulation, card games, and scenario simulation. We hope this research will help us understand whether this new model can more effectively help you master the knowledge and skills of internal medicine nursing, and cultivate clinical thinking abilities and learning interest.

## 2. What Will You Need to Do?

If you agree to participate, you will be invited to take part in this study:

This study will last for one semester, concurrent with your Internal Medicine Nursing practical course.

You will be randomly assigned to either an "Experimental Group" or a "Control Group."

The Experimental Group will experience the new blended teaching model, including using an AI learning assistant, participating in card-based desktop exercise games, scenario simulation practices, etc.

The Control Group will undergo learning according to the existing traditional teaching methods.

All teaching activities are regular components of the Internal Medicine Nursing course and will not occupy your additional rest time.

During the study, we will collect some data for analysis, including:

Your course scores (theoretical exam and practical skill assessment scores).

Anonymous teaching satisfaction questionnaires you complete.

(For some students in the Experimental Group only) We might invite you to participate in an anonymous interview lasting approximately 20-30 minutes to share your learning experiences and feelings. The interview content will be audio-recorded and transcribed for analysis, but your personal information will be kept strictly confidential.

#### 3. Potential Risks and Discomforts

The risks associated with participating in this study are minimal. All teaching activities fall within the regular teaching plan. The interview might take up some of your extracurricular time, and you are free to choose whether or not to participate. If you feel any discomfort during participation, you can pause or withdraw at any time.

#### 4. Potential Benefits

You may not receive direct personal benefits from this study. However, your participation will provide us with valuable information to help improve future teaching methods, benefiting your junior fellow students and contributing to the development of nursing education.

# 5. Confidentiality

Your privacy will be protected at the highest level:

All collected data (scores, questionnaires, interview records) will be anonymized. Your name will be replaced by a unique code.

All research data will be encrypted and stored on secure servers, accessible only to authorized members of the research team.

No personally identifiable information will appear in the final research report or any publications.

# 6. Voluntary Participation and Right to Withdraw

Your participation is entirely voluntary.

You have the right to refuse to participate in this study, which will not negatively affect your academic grades, teacher-student relationship, or any rights you enjoy at the university.

Even after signing this consent form, you can choose to withdraw from the study at any time, without providing any reason, and without any adverse consequences.

#### 7. Contact Information

If you have any questions, concerns, or encounter any problems during the research process, please feel free to contact the principal researcher using the contact information provided above.

## Participant Statement

Date: Month Day, Year

I have read and understood the above information about this study. I have had the opportunity to ask questions and have received satisfactory answers. I voluntarily agree to participate in this research.

| I understand that I can withdraw at any time without penalty | • |
|--------------------------------------------------------------|---|
| Participant Name (Printed): | |
| Participant Signature: | |

| Researcher S | Statement |
|--------------|-----------|
|--------------|-----------|

| I confirm that I have explained the purpose, procedures, and precautions of this study to the participant and have answered all their questions. |
|---|
| Researcher Signature: |
| Date: Month Day, Year |